CLINICAL TRIAL: NCT06468943
Title: Polatuzumab Vedotin and Zanubrutinib Plus R-CHP for Patients in Treatment of Newly Diagnosed Untreated Non-GCB DLBCL With Extranodal Involvement.
Brief Title: Polatuzumab Vedotin and Zanubrutinib Plus R-CHP for Patients With Newly Diagnosed Untreated Non-GCB DLBCL
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pola-ZR-CHP
Record Dates: First submitted 2024-04-27; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-04

CONDITIONS: Effects of Chemotherapy; Safety Issues
MeSH Terms: interventions — polatuzumab vedotin; zanubrutinib; Rituximab; Cyclophosphamide; Doxorubicin; Prednisone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients receiving Pola+ZR-CHP treatment (Experimental)
  Interventions: Drug: Polatuzumab Vedotin; Drug: Zanubrutinib; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Prednisone

INTERVENTIONS:
Drug: Polatuzumab Vedotin — 1.8mg/kg/21d（d0） Intravenous infusion
Drug: Zanubrutinib — 160mg bid PO（d0-d20）
Drug: Rituximab — 375mg/㎡/21d（d0） Intravenous infusion
Drug: Cyclophosphamide — 750mg/㎡/21d（d1） Intravenous infusion
Drug: Doxorubicin — 50mg/㎡/21d（d1） Intravenous infusion
Drug: Prednisone — 100mg PO （d1-d5）/21d

SUMMARY:
Aim of this study will evaluate the efficacy and safety of Polatuzumab Vedotin and Zanubrutinib in combination with R-CHP for newly diagnosed untreated Non-GCB DLBCL Patients with extranodal involvement.

DETAILED DESCRIPTION:
Diffuse large B-cell lymphoma (DLBCL) is the most common type of non-Hodgkin's lymphoma. According to Hans' algorithms, DLBCL can be identified as 2 subtypes: germinal b-cell-like(GCB) and non-germinal b-cell-like(non-GCB). Approximately 50 to 60% of DLBCL was non-GCB subtype DLBCL.The non-GCB DLBCL revealed poor clinical outcomes. Bruton's tyrosine kinase (BTK) inhibitors have established therapeutic activity in B cell malignancies, with potential activity in non-GCB DLBCL. The POLARIX study also observed an benefit in the efficacy of Polatuzumab Vedotin in first-line treatment of DLBCL patients. This study will evaluate the efficacy and safety of Polatuzumab Vedotin and Zanubrutinib in combination with R-CHP for newly diagnosed untreated Non-GCB DLBCL Patients with extranodal involvement.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed Non-GCB DLBCL with extrinsic involvement；
2. Measurable disease of at least 15mm(node)/10mm（extranodal）；
3. ECOG performance status 0-2；
4. Adequate organ function:Cardiac ejection fraction (EF) ≥ 50%;Creatinine clearance rate (≥30 mL/min) of serum creatinine; Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) ≤3 times ULN；
5. Adequate bone marrow function:Platelet count (≥ 50×10^9/L);Hemoglobin (≥ 8 g/dL);The absolute value of neutrophils (≥1.0×10^9/L)
6. Estimated survival time ≥3 months
7. Subjects of child-bearing or child-fathering potential must be willing to practice birth control from the time of enrollment on this study until the follow-up period of the study.

Exclusion Criteria:

1. Accepted major surgery within 4 weeks before treatment;
2. Diagnosis of primary mediastinal lymphoma or primary CNS lymphoma;
3. Previous history of indolent lymphoma;
4. Prior malignancy (other than DLBCL), except for cured malignant tumors with no active lesions for 3 years;Adequate treatment of inactive lesions in non-melanoma skin cancer 、malignant tonsilloma or carcinoma in situ;
5. History of intracranial haemorrhage in preceding 6 months,requires or receiving anticoagulation with warfarin or equivalent antagonists;
6. Requires treatment with a strong/medium CYP3A inducer;
7. The previous use of anthracycline-based drugs > 150 mg/m2;
8. Evidence of complications or medical conditions, including but not limited, that may interfere the conduct of the study or place the patient at serious risk:significant cardiovascular disease(class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification、myocardial infarction within 6 months of screening、uncontrolled or symptomatic arrhythmias) and/or significant lung disease;
9. HIV infection and/or active hepatitis B or active hepatitis C;
10. Uncontrolled systemic infection;
11. Pregnant or breasting-feeding women;
12. According to the researchers' judgment, patients' underlying condition may increase their risk of receiving research drug treatment, or confuse their judgment on toxic reactions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival（PFS） | From date of enrollment until the date follow up for 2 years after the treatment or progression disease or date of death for any cause.
  The time between enrollment and tumor occurrence (in any aspect) progression or (for any reason) death

SECONDARY OUTCOMES:
Objective Response rate（ORR） | From date of enrollment until the date follow up for 2 years after the treatment or progression disease or date of death for any cause.
  The proportion of patients who achieved complete or partial response in efficacy evaluation at the end of treatment
Complete Response（CR） | From date of enrollment until the date follow up for 2 years after the treatment or progression disease or date of death for any cause.
  The proportion of patients who achieved complete response in efficacy evaluation at the end of treatment
Duration of Response（DOR） | All time in the study
  It refers to the time from the first assessment of a tumor as CR or PR to the second assessment as PD (Progressive Disease) or death from any cause.
Overall Survival | From date of enrollment until the date follow up for 2 years after the treatment or progression disease or date of death for any cause.
  The time between enrollment to death(for any reason) .
Adverse Events(AEs) | From date of enrollment until the date follow up for 2 years after the treatment or progression disease or date of death for any cause.
  All treatment-related adverse events that occur during patient treatment and follow-up.

OTHER OUTCOMES:
Exploratory study endpoint | From date of enrollment until the date follow up for 2 years after the treatment or progression disease or date of death for any cause.
  Exploring the therapeutic response of subjects with different genotypes to Pola+ZR-CHP regimen using Next-generation sequencing(NGS).

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Nanjing, China